CLINICAL TRIAL: NCT06176742
Title: Comparative Effects of Active Cycle Breathing Technique and Bubble Positive Expiratory Pressure Device in Asthmatic Patients
Brief Title: Comparative Effects of ACBT and Bubble Positive Expiratory Pressure Device in Asthmatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0330
Record Dates: First submitted 2023-10-26; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Asthma
Keywords: Asthma; Active Cycle Breathing Technique; Bubble PEP
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bubble Positive Expiratory Pressure Device (Experimental): Diaphragmatic breathing technique will be the baseline treatment. B group will be treated with bubble positive expiratory pressure device. Patients will be encouraged to blow down the tubing into the water, and make bubbles. This creates positive pressure back up the tubing and into patient's airways and lungs. As the pressure holds open your patient's airways, it helps more air to move in and out of their lungs. All study participant will receive a total of 18 treatment sessions over a six-week period, which consisted of 03 treatment sessions per week.
  Interventions: Other: Bubble Positive Expiratory Pressure Device
- Active Cycle Breathing Technique (Active Comparator): Diaphragmatic breathing technique will be the baseline treatment.A group will be treated with active cycle breathing technique. The technique consists of inspiratory hold technique, deep breathing and forced expiration. These are repeated in a cycle until your chest feels clear. You can carry out ACBT when either sitting or lying down.
  Physiotherapist will discuss this with you during your physiotherapy assessment. All study participant will receive a total of 18 treatment sessions over a six-week period, which consisted of 03 treatment sessions per week.
  Interventions: Other: Active Cycle Breathing Technique

INTERVENTIONS:
Other: Active Cycle Breathing Technique — This study will be Randomized Clinical trial, Subject diagnosed with asthma meeting predetermined inclusion and exclusion criteria and will be divided into two groups. The baseline treatment for both groups would be diaphragmatic breathing exercises. While group A will be treated with ACBT. Each subject will receive 18 sessions with 3 treatments per week. Post treatment values will be recorded after the session and recorded values will be analyzed using SPSS 25.
  Arms: Active Cycle Breathing Technique
Other: Bubble Positive Expiratory Pressure Device — This study will be Randomized Clinical trial, Subject diagnosed with asthma meeting predetermined inclusion and exclusion criteria and will be divided into two groups. The baseline treatment for both groups would be diaphragmatic breathing exercises. While group B will be treated with bubble-PEP. Each subject will receive 18 sessions with 3 treatments per week. Post treatment values will be recorded after the session and recorded values will be analyzed using SPSS 25.
  Arms: Bubble Positive Expiratory Pressure Device

SUMMARY:
The study gap is that in previous studies the effects of bubble-PEP in different diseases have been studied but it's never been studied in asthmatic patients, so the reason behind this study is to see effects of bubble-PEP in Asthmatic Patients.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of Bubble-PEP device compared to ACBT in asthmatic patients. This study will be Randomized Clinical trial, Subject diagnosed with asthma meeting predetermined inclusion and exclusion criteria and will be divided into two groups. The baseline treatment for both groups would be diaphragmatic breathing exercises. While group A will be treated with ACBT and group B will be treated with bubble-PEP device. Each subject will receive 18 sessions with 3 treatments per week. Post treatment values will be recorded after the session and recorded values will be analyzed using SPSS 25

ELIGIBILITY:
Inclusion Criteria:

* Aged between 31 to 40 years
* Male & Female
* Mild Asthmatic Patients
* Able to perform techniques
* Those who have never taken therapies for asthma before.
* Chronic Asthma

Exclusion Criteria:

* Patients with hypertension
* Cardiac diseases
* Any rib fracture
* Previously taken instructions regarding this.
* Any other unstable medical conditions

Ages: 31 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Dyspnea 12 Tool | Up to 24 weeks
  Dyspnea 12 is a valid and reliable measure of breathlessness in patients. It measures the current level of a patients breathlessness severity, incorporating both physical and affective aspects and does not depend on activity limitation. D-12 consists of 12 descriptor items on a scale of none (0), mild (1), moderate (2), or severe (3). It provides an overall score for breathlessness severity that incorporates seven physical items and five affective items. The time reference period captures the current level of breathlessness experienced by patients as opposed to specifically on the day of the test or in response to a specific activity. Data will be calculated before and after treatment with the help of outcome measure tools.
Breathlessness, Cough, and Sputum Scale (BCSS) | Upto 24 weeks
  The breathlessness, cough and sputum scale (BCSS) is used to predict patient exacerbation by evaluating common symptoms. The BCSS tool measures the patients self reported symptoms in real time. BCSS is a patient-reported outcome measure that asks patients to rate the severity of the three symptoms, each on a 5-point scale; from 0 to 4 the higher scores indicate more severe symptoms. Item scores are summed to yield a total score. Data will be calculated before and after treatment with the help of outcome measure tools.
Pulmonary Function Test | Upto 24 weeks
  Pulmonary function tests measure how much air you can exhale, and how quickly. There are several types of pulmonary function graphs that show data from the tests. The test which will be used is FEV1/FVC. This is the amount of air exhaled in the first second, compared with the total amount of air exhaled. It's given as a fraction (ratio) or a percentage. In general, the higher the FEV1/FVC, the better. This test will be done using Spirometer. Data will be calculated before and after treatment with the help of outcome measure tools.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Altaf, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Muzaffargarh, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santos MD, Milross MA, McKenzie DK, Alison JA. Bubble-positive expiratory pressure device and sputum clearance in bronchiectasis: A randomised cross-over study. Physiother Res Int. 2020 Jul;25(3):e1836. doi: 10.1002/pri.1836. Epub 2020 Feb 29. PMID 32113192
- [Background] Phillips J, Hing W, Pope R, Canov A, Harley N, Lee AL. Active cycle of breathing technique versus oscillating PEP therapy versus walking with huffing during an acute exacerbation of bronchiectasis: a randomised, controlled trial protocol. BMC Pulm Med. 2023 Jan 25;23(1):36. doi: 10.1186/s12890-023-02324-8. PMID 36698169
- [Background] Mestriner RG, Fernandes RO, Steffen LC, Donadio MV. Optimum design parameters for a therapist-constructed positive-expiratory-pressure therapy bottle device. Respir Care. 2009 Apr;54(4):504-8. PMID 19327187
- [Background] Sehlin M, Ohberg F, Johansson G, Winso O. Physiological responses to positive expiratory pressure breathing: a comparison of the PEP bottle and the PEP mask. Respir Care. 2007 Aug;52(8):1000-5. PMID 17650355
- [Background] Lewis LK, Williams MT, Olds TS. The active cycle of breathing technique: a systematic review and meta-analysis. Respir Med. 2012 Feb;106(2):155-72. doi: 10.1016/j.rmed.2011.10.014. Epub 2011 Nov 18. PMID 22100537
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Chanez P, Wenzel SE, Anderson GP, Anto JM, Bel EH, Boulet LP, Brightling CE, Busse WW, Castro M, Dahlen B, Dahlen SE, Fabbri LM, Holgate ST, Humbert M, Gaga M, Joos GF, Levy B, Rabe KF, Sterk PJ, Wilson SJ, Vachier I. Severe asthma in adults: what are the important questions? J Allergy Clin Immunol. 2007 Jun;119(6):1337-48. doi: 10.1016/j.jaci.2006.11.702. Epub 2007 Apr 9. PMID 17416409
- [Background] Bousquet J, Mantzouranis E, Cruz AA, Ait-Khaled N, Baena-Cagnani CE, Bleecker ER, Brightling CE, Burney P, Bush A, Busse WW, Casale TB, Chan-Yeung M, Chen R, Chowdhury B, Chung KF, Dahl R, Drazen JM, Fabbri LM, Holgate ST, Kauffmann F, Haahtela T, Khaltaev N, Kiley JP, Masjedi MR, Mohammad Y, O'Byrne P, Partridge MR, Rabe KF, Togias A, van Weel C, Wenzel S, Zhong N, Zuberbier T. Uniform definition of asthma severity, control, and exacerbations: document presented for the World Health Organization Consultation on Severe Asthma. J Allergy Clin Immunol. 2010 Nov;126(5):926-38. doi: 10.1016/j.jaci.2010.07.019. PMID 20926125
- [Background] Wenzel SE. Asthma: defining of the persistent adult phenotypes. Lancet. 2006 Aug 26;368(9537):804-13. doi: 10.1016/S0140-6736(06)69290-8. PMID 16935691
- [Background] Murphy AC, Proeschal A, Brightling CE, Wardlaw AJ, Pavord I, Bradding P, Green RH. The relationship between clinical outcomes and medication adherence in difficult-to-control asthma. Thorax. 2012 Aug;67(8):751-3. doi: 10.1136/thoraxjnl-2011-201096. Epub 2012 Mar 21. PMID 22436168
- [Background] Mahdaviani SA, Rezaei N, Moradi B, Dorkhosh S, Amirzargar AA, Movahedi M. Proinflammatory cytokine gene polymorphisms among Iranian patients with asthma. J Clin Immunol. 2009 Jan;29(1):57-62. doi: 10.1007/s10875-008-9232-1. Epub 2008 Sep 2. PMID 18763028
- [Background] Bousquet J, Dahl R, Khaltaev N. Global alliance against chronic respiratory diseases. Allergy. 2007 Mar;62(3):216-23. doi: 10.1111/j.1398-9995.2007.01307.x. PMID 17298337
- [Background] Zuriati Z, Surya M. Effectiveness Active Cycle of Breathing Technique (ACBT) with Pursed Lips Breathing Technique (PLBT) to tripod position in increase oxygen saturation in patients with COPD, West Sumatera. Enfermeria Clinica. 2020 Jun 1;30:164-7.
- [Background] Eastwood B, Jepsen N, Coulter K, Wong C, Zeng I. Challenges of undertaking a clinical trial using bubble-PEP in an acute exacerbation of chronic obstructive pulmonary disease: A feasibility study. New Zealand Journal of Physiotherapy. 2016 Mar 1;44(1).
- [Background] Sundus S, Memoona S, Muhammad IN, Rashid HN. Effect of Active Cycle of Breathing Technique in Adult Asthmatic Patients in Pakistan. Asian Journal of Medicine and Biomedicine. 2017 Dec 21;1(1):32-